CLINICAL TRIAL: NCT05133284
Title: Evaluation of the Effectiveness of the Therapeutic Education Program "Living Better With ADHD" in Improving the Quality of Life of Children With ADHD and Their Parents
Brief Title: Effectiveness of a Therapeutic Education Program in Improving Quality of Life of Children With ADHD and Their Parents
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0634
Record Dates: First submitted 2021-10-22; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-10

CONDITIONS: Attention Deficit Disorder
Keywords: Therapeutic Education; Quality of life
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Attention Deficit Hyperactivity Disorder (ADHD) is a neurodevelopmental disorder characterized by attention deficit, impulsivity and hyperactivity. It's one of the most frequently encoutered disorder in child psychiatry. ADHD has a significant impact on the quality of life of children and their parents.

In the child psychiatry department of the MPEA Peyre Plantade, a Therapeutic Education program specific to ADHD has been set up for children and their parents. This program consists of different workshops whose aim is to reduce the ADHD repercussions on the daily life of children and their families and thus improve their quality of life.

The principal aim of our study is to evaluate the effectiveness of this program in improving the quality of life of children with ADHD and their parents.

ELIGIBILITY:
Inclusion criteria:

* Aged 8 to 13
* With a diagnosis of ADHD
* Living in the herault department
* Participatinf in the therapeutic education program " Living Well with ADHD "

Exclusion criteria:

* Parent's objection to the use of data collected
* Parent unable to complete questionnaires

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and adolescents, aged 8 to 13, with a diagnosis of ADHD and participating in the therapeutic education program " Living Well with ADHD "
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-25 (Estimated)

PRIMARY OUTCOMES:
Quality of life of children | 1 day
  To Evaluate the effectiveness of the therapeutic education program "Living better with ADHD" in improving quality of life of children with ADHD measured by the Kidscreen 27 questionnaire (Total score & sub score)

OTHER OUTCOMES:
Quality of life of parents | day 1
  To evaluate the effectiveness of the program in improving the overall quality of life of parents measured by the WHOQOL-BREF questionnaire (Total score & sub score)
Clinical and sociodemiographic characteristics | day 1
  To Identify Clinical and sociodemographic characteristics that influence the quality of life of children and parents

CONTACTS AND LOCATIONS:
Overall Officials: Amaria BAGHDADLI, PU-PH, Study Director — University Hospital, Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC